CLINICAL TRIAL: NCT02402192
Title: A Prospective Randomized Trial to Analyze the Effect of the Gonadotropin Administered During Control Ovarian Stimulation on Embryo Kinetics of Development
Brief Title: Type of Gonadotropin and Embryo Kinetics of Development
Acronym: PEM-ESD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, PhD MD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411-MAD-079-CB
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Infertility
Keywords: corifollitropin alfa; recombinant FSH; HP-hMG; time-lapse; kinetics of development
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Corifollitropin alfa (Active Comparator): Under current practice, 67 participants will be stimulated with a single injection of 100 mg, sc of Corifollitropin alpha (Elonva®). From day 6 stimulation and even prior to induction of ovulation day, 0.25 mg / day was administered sc ganirelix (Orgalutran®). From day 8 stimulation and depending on the ovarian response, you can add recombinant FSH (Puregon) up to 150 IU by Puregon Pen® device. In the presence of 3 or more follicles ≥17 mm, ovulation is induced with a single dose of 0.2 mg Decapeptyl 6500u or hCG (Ovitrelle) if there is no risk of OHSS, and 36 hours later he held the follicular puncture oocyte retrieval.
  Interventions: Drug: Corifollitropin alfa
- recombinant FSH (Active Comparator): Under current practice, 67 participants will be stimulated with a daily dose of recombinant FSH. Administration of recombinant FSH (Puregon) starts at an initial dose of 150-225 IU / day by the Puregon Pen® device. From day 6 stimulation 0.25 mg / day administered sc ganirelix (Orgalutran®). From this day may also vary the dose of recombinant FSH according ovarian response. In the presence of 3 or more follicles ≥17 mm, a single dose of 0.2 mg or Decapeptyl hCG 6500u (Ovitrelle) is given if there is no risk of OHSS, and 36 hours then held follicular puncture for recovering oocytes.
  Interventions: Drug: Corifollitropin alfa
- HP- hMG (Active Comparator): Under current practice, 67 participants will be stimulated with HP-hMG, following the same pattern described for the group of recombinant FSH. In this case, the initial dose is 225-300 IU / day of HP-hMG (Menopur®). From day 6 stimulation 0.25 mg / day administered sc ganirelix (Orgalutran®). From this day may also vary the dose of HP-hMG according ovarian response. In the presence of 3 or more follicles ≥17 mm, a single dose of 0.2 mg Decapeptyl 6500u or hCG (Ovitrelle) is given if there is no risk of OHSS and 36 hours then held the follicular puncture for oocyte retrieval .
  Interventions: Drug: Corifollitropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa
  Other Names: Elonva

SUMMARY:
The study is proposed to determine the effect of three types of gonadotropins that are currently used in protocols of controlled ovarian stimulation in women undergoing in vitro fertilization techniques on the kinetics of embryonic development.

ELIGIBILITY:
Inclusion Criteria:

* Women <38 years old
* Weight <60 kg
* Own oocytes
* Patients have to provide signed informed consent

Exclusion Criteria:

* Oocyte donors
* Vitrified oocytes
* Severe male factor (<1 million spz/ml)
* Weight >60 kg

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
T5 defined as the time that embryo needs to reach a 5-cell stage. | Baseline

SECONDARY OUTCOMES:
Length of stimulation (days) | a month
Total dose of gonadotropins (IU) | A month
Levels of FSH (IU) Levels of estradiol (pg / ml) - Levels of progesterone (ng / ml) - Fertilization rate - Number of embryos transferred and cryopreserved - Pregnancy rate - Implantation | A month
Levels of estradiol (pg / ml) Number of embryos transferred and cryopreserved - Pregnancy rate - Implantation | A month
Levels of progesterone (ng/ml) | A month
Fertilization rate | A month
Number of embryos transferred and cryopreserved | A month
Pregnancy rate | A month
Implantation rate | A monthe
Miscarriage rate | A month
Cancellation rate per cycle initiated | A month
Ovarian hyperstimulation syndrome rate | A month
Timings of cellular divisions | A month

REFERENCES:
- [Background] Meseguer M, Rubio I, Cruz M, Basile N, Marcos J, Requena A. Embryo incubation and selection in a time-lapse monitoring system improves pregnancy outcome compared with a standard incubator: a retrospective cohort study. Fertil Steril. 2012 Dec;98(6):1481-9.e10. doi: 10.1016/j.fertnstert.2012.08.016. Epub 2012 Sep 10. PMID 22975113
- [Result] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043
- [Result] Garcia-Velasco JA, Zuniga A, Pacheco A, Gomez R, Simon C, Remohi J, Pellicer A. Coasting acts through downregulation of VEGF gene expression and protein secretion. Hum Reprod. 2004 Jul;19(7):1530-8. doi: 10.1093/humrep/deh298. Epub 2004 May 20. PMID 15155606
- [Result] Requena A, Cruz M, Collado D, Izquierdo A, Ballesteros A, Munoz M, Garcia-Velasco JA. Evaluation of the degree of satisfaction in oocyte donors using sustained-release FSH corifollitropin alpha. Reprod Biomed Online. 2013 Mar;26(3):253-9. doi: 10.1016/j.rbmo.2012.11.015. Epub 2012 Dec 5. PMID 23352098
- [Result] Seyhan A, Ata B. The role of corifollitropin alfa in controlled ovarian stimulation for IVF in combination with GnRH antagonist. Int J Womens Health. 2011;3:243-55. doi: 10.2147/IJWH.S15002. Epub 2011 Aug 8. PMID 21892335
- [Result] Meseguer M, Herrero J, Tejera A, Hilligsoe KM, Ramsing NB, Remohi J. The use of morphokinetics as a predictor of embryo implantation. Hum Reprod. 2011 Oct;26(10):2658-71. doi: 10.1093/humrep/der256. Epub 2011 Aug 9. PMID 21828117